CLINICAL TRIAL: NCT04578951
Title: Measurement of the Quality of Life in Patients Operated With a Total Knee Prosthesis (TKA) From the FHK® Range and Followed for 2 Years.
Brief Title: Measurement of the Quality of Life in Patients Operated With a Total Knee Prosthesis (TKA) From the FHK® Range.
Status: Terminated | Type: Observational
Why Stopped: Only 19% of the expected patients have been enroled. Patient's follow-up has not been realized as expected in the protocol
Sponsor: FH ORTHO (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-41
Record Dates: First submitted 2020-09-22; First posted 2020-10-08 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Knee Disease
Keywords: Knee; Arthroplasty; Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients receiving a prosthesis from the FHK® range
  Interventions: Device: FHK® total knee prosthesis

INTERVENTIONS:
Device: FHK® total knee prosthesis — FHK® prosthesis are intended to be implanted in the tibial and femoral regions during total knee arthroplasty in order to restore joint function.

SUMMARY:
As part of Medical Devices CE marking regulatory process, an appropriate post-market clinical follow-up (PMCF) is required. This PMCF study is in the framework of CE mark renew of FHK® total knee prosthesis, it aims to answer specific questions related to safety and performance of the device, when used in accordance with the approved instructions for use.

This study is based on a quality of life self-assessment from the preoperative to postoperative phases and up to two years of follow-up.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the quality of life in patients operated with a FHK® total knee prosthesis up to 2 years of follow-up.

The secondary objectives are to evaluate the security and performance of the devices by gathering complications, revision rate of the devices (survival analysis) and functional score up to 2 years of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subject implanted with FHK® prosthesis in one of the following indication according to the instructions for use: knee disorders; Aseptic condylar necrosis.
* Subject who received an information form and is willing to participate in the study.
* Adults subjects (≥18 years old).
* Access to an internet connection allowing to complete the questionnaires on the online platform

Exclusion Criteria:

* Contraindications described in the instructions for use
* Subject who is not able to express his/her non-opposition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from participating hospitals will be enrolled as part of their clinical routine care
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Quality of life EQ-5D-5L score | 14 days preoperative ; 70 days post-op, 177 days post-op, 357 days post-op, 717 days post-op
  The primary outcome measures will be determined by the EQ-5D-5L score. The EQ-5D-5L score is a self-administered quality of life questionnaire by patients. The EQ-5D-5L consists of two parts, One part with a five-dimensional system and the last one is a visual analog scale graduated from 0 to 100. We will observe the evolution of this score according to the time frame.

SECONDARY OUTCOMES:
Survival rate | 2 years post-op
Evolution of parameters describing pain, stability, knee mobility and patient autonomy | From the preoperative visit to 2 years postoperative.
  The secondary outcome measures will be determined by the KOOS-PS score, a patellar evaluation, and questions about physical abilities.
  The KOOS-PS score is a score used in the clinical evaluation of various knee pathologies.This score assesses both the long and medium term consequences of a knee injury. It contains 42 items in 5 separately scored subscales (pain, other symptoms, function in daily life, function in leisure and sports and quality of life related to the knee).
  The patellar evaluation is a questionnaire assessing the functional state of the knee with questions such as the level of pain in the anterior region of the knee, assessment of the strength of the quadriceps, the ability to rise from a chair.
  Physical abilities will be assessed with questions like the patient's walking distance, the ability to cycle, the ability to go shopping.
Rate of complications | All complications will be gathered during intervention and up to 2 years postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique du Maine, Laval, France

IPD SHARING:
Plan to Share IPD: No